CLINICAL TRIAL: NCT00834236
Title: Diagnosis of Gastroduodenal Diseases by Proteiomic Fingerprints of Gastric Juice
Brief Title: Proteiomic Fingerprints of Gastric Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VGHKS96-CT2-24
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; proteomics; gastric juice
MeSH Terms: conditions — Stomach Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gastric cancer (Experimental): gastric cancer patients
  Interventions: Other: normal subject; Other: gastric cancer
- normal subject (Active Comparator): healthy subject
  Interventions: Other: normal subject; Other: gastric cancer

INTERVENTIONS:
Other: normal subject — biomarker in gastric juice, i.e., alpha 1-antitrypsin, CEA
  Other Names: biomarker in gastric juice
Other: gastric cancer — biomarker in gastric juice, e.g., alpha 1-antitrypsin
  Other Names: biomarker in gastric juice

SUMMARY:
No accurate, inexpensive and non-invasive test for gastric cancer screening is currently available. The investigators' recent study identified a1-antitrypsin and other proteins as potential biomarkers of gastric cancer in gastric juice. The aim of this study was to develop a novel non-invasive modality for detecting gastric cancer by measurement of biomarkers in gastric juice.

DETAILED DESCRIPTION:
Patients and methods: The study consisted of two parts: (1) investigating the differences in gastric juice biomarker concentrations between gastric cancer patients and controls, and (2) screening gastric cancer using string test to obtain gastric juice followed by immunoassay for biomarker concentration.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects and gastric cancer patients documented by endoscopy.

Exclusion Criteria:

* the use of proton pump inhibitors or histamine-2 receptor antagonists within 4 weeks prior to the study
* coexistence of two kinds of gastroduodenal lesions
* coexistence of severe systemic diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, M.D., Principal Investigator — Kaohsiung Veterans Genaral hospital
Locations (2):
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung
  - Kaohsiung Veterans General Hospital, Kaohsiung City

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gastric Cancer | Normal Subject
Started | 29 | 47
Completed | 29 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Cancer | Normal Subject | Total
Number analyzed (Participants) | 29 | 47 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 42 | 52
  >=65 years | 19 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (14.3) | 51.4 (14.9) | 59.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 33
  Male | 20 | 23 | 43
Region of Enrollment [Number; unit: participants]
  Taiwan | 29 | 47 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate Diagnosis for Gastric Cancer
Description: Normal subject group: number of the subjects with normal alpha 1-antitrypsin level in gastric juice Gastric cancer group: number of the subjects with elevated alpha 1-antitrypsin level in gastric juice
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Gastric Cancer | Normal Subject
Number analyzed (Participants) | 29 | 47
participants | 27 | 44

ADVERSE EVENTS:
Arm/Group | Gastric Cancer | Normal Subject
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/47
Other Adverse Events (participants affected / at risk) | 0/29 | 0/47

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes